CLINICAL TRIAL: NCT01530230
Title: Randomised Study on Cardiac Effects of Oxytocin During Caesarean Section in Preeclamptic Women
Brief Title: ST- Depression on Electrocardiogram During Caesarean Section in Regional Anaesthesia in Women With Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Maria Jonsson, Principal investigator, Uppsala University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 2004-74
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Preeclampsia
Keywords: cesarean section; electrocardiography; heart; hypotension; ischemia; oxytocin; preeclampsia; regional anesthesia; ECG changes suggestive of myocardial ischemia
MeSH Terms: conditions — Pre-Eclampsia; Hypotension; Ischemia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Oxytocin 5 units (Other)
  Interventions: Drug: oxytocin
- Oxytocin 10 units (Other)
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — Intravenous bolus dose given during 1 minute after clamping of the umbilical cord

SUMMARY:
The investigators examined whether there was a difference in the occurrence of ST depressions after injection of five or ten units of oxytocin, in preeclamptic patients delivered by caesarean section (CS) under regional anesthesia.

DETAILED DESCRIPTION:
ST depression on electrocardiograms has been reported in healthy women undergoing cesarean section in regional anesthesia. The investigators examined whether there was a difference in the occurrence of electrocardiogram changes suggestive of myocardial ischemia (ST depressions) in preeclamptic patients randomized to five or ten units of oxytocin during cesarean section with regional anesthesia.

In a double-blind randomized controlled study preeclamptic patients undergoing cesarean section under spinal anesthesia were randomized to 5 or 10 units of oxytocin, given as an intravenous bolus. A Holter monitor was used to record electrocardiograms. Non-invasive blood pressure and heart rate were monitored.

ELIGIBILITY:
Inclusion Criteria:

* women with preeclampsia undergoing CS under spinal anesthesia. Preeclampsia was diagnosed if blood pressure was ≥ 140/90 mm Hg and if proteinuria of more than 1000 mg/day persisted.

Exclusion Criteria:

* multiple birth,
* obesity (body mass index > 35),
* age < 18 years,
* complications of the pregnancy other than preeclampsia or non-proficiency in the Swedish language

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Depression of the ST segment on electrocardiograms | From start of caesarean section until 20 minutes after delivery

SECONDARY OUTCOMES:
Mean arterial pressure and heart rate. | From start of caesarean section until 20 minutes after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obsterics and Gynecology, Uppsala, Sweden